CLINICAL TRIAL: NCT04271033
Title: Long-term Outcomes of MicroNet-covered Stent Routine Use for Stroke Prevention in Symptomatic and Increased-risk Asymptomatic Carotid Stenosis Patients Requiring Revascularization by Neurovascular Team Decision: PARADIGM-EXTEND
Brief Title: MicroNet-covered Stent System for Stroke Prevention in All Comer Carotid Revascularization
Acronym: PARADIGM-EXT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: John Paul II Hospital, Krakow (Other)
Collaborators: Jagiellonian University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PARADIGM-EXTEND
Record Dates: First submitted 2020-01-15; First posted 2020-02-17 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Carotid Artery Diseases
Keywords: Stenting
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Intervention Model Description: Single arm registry
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carotid Artery Stenting (Experimental): Consecutive male and female patients older than 18 year with symptomatic and increased-stroke-risk asymptomatic carotid lesions that require revascularization by Neurovascular Team decision.
  Interventions: Device: Carotid Artery Stenting

INTERVENTIONS:
Device: Carotid Artery Stenting — Carotid artery stenting according to local clinical experience and ESC/ESVS guidelines using exclusively CGuard™, MicroNet covered stent under proximal or distal intraprocedural cerebral protection according to "tailored CAS" algorithm.

SUMMARY:
All-comer study of unselected patients suitable for carotid artery revascularization to evaluate the feasibility, efficacy and safety of first line endovascular revasculariztion using MicroNet covered stent (CGuard™) in the treatment of consecutive symptomatic and increased-stroke-risk asymptomatic carotid lesions that require revascularization by Neurovascular Team decision.

DETAILED DESCRIPTION:
Independent investigator initiated, academic, single arm, open-label, non-randomized, prospective, multicenter, multispecialty trial of CGuard™ routine use in all-comer population of consecutive patients with symptomatic or increased-stroke-risk asymptomatic carotid stenosis.

Increased-stroke-risk is defined as the following patient and/or lesion characteristics:

thrombus containing, documented progressive, irregular, ulcerated lesion; evidence of ipsilateral ischemic cerebral injury in MRI or CT imaging; contralateral stroke in relation to carotid stenosis; contralateral artery occlusion.

The main objective of this observational study is to evaluate (1) the periprocedural feasibility and efficacy of CGuard™ stent system in the treatment of carotid artery stenosis (2) long-term efficacy and safety of routine CGuard™ stent system use.

The study hypothesis is that the novel CGuard™ MicroNet® covered stent is safe and effective for a majority of consecutive patients considered to require carotid revascularization.

The multicenter arm of the project has a specific cohort descriptor: PARADIGM-EXTEND MC

ELIGIBILITY:
General Inclusion Criteria:

* Patient > 18 years old qualified by NeuroVascular Team for carotid revascularization according to local standards of care
* Signed informed consent
* Agreement (routin un this group of patients) to clinical and ultrasonographis follow up.

Angiographic Inclusion Criteria:

* De-novo atherosclerotic lesions or neo-atherosclerosis
* Symptomatic patients (history of transient ischemic attack, ischaemic stroke or amaurosis fugax within 6 months from index procedure) with index artery stenosis ≥50% assessed in angiography with NASCET method or
* Asymptomatic patients with index artery stenosis ≥70-80% assessed in angiography with NASCET method

General Exclusion Criteria:

* Lack of NeuroVascular Team agreement on carotid revascularization indication
* Lack of signed informed consent
* Estimated life expectancy less than 1 year
* Chronic renal failure with serum creatinine level > 3.0 mg/dL
* Myocardial Infarction within 72 hours prior to index procedure.
* Pregnant women
* Diagnosed coagulopathies
* History of contrast media allergy, not reacting to pharmacotherapy

Angiographic Exclusion Criteria:

* Index lesion occlusion
* Common carotid artery stent protruding to aortic arch
* Anatomical conditions restricting stent implantation
* Significant common carotid artery stenosis proximal to index lesion (unless treated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2015-09-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
MACNE (Major Adverse Cardiac and Neurological Events) | 12 months
  Death, Stroke, Myocardial Infarction.

SECONDARY OUTCOMES:
Procedural success | Within 48 hours from index procedure
  Successful stent delivery and deployment without complication
In-hospital MACNE (Major Adverse Cardiac and Neurological Events) | Within 48 hours from index procedure
  Death, Stroke, Myocardial Infarction within index hospitalization
30-day MACNE (Major Adverse Cardiac and Neurological Events) | 30 days
  Death, Stroke, Myocardial Infarction within 30 days
Incidence of any periprocedural complications | Within 48 hours
  Any periprocedural complications
Functional MRI efficacy assessment. | Within 48 hours
  In case of fMRI evaluation, pre and postprocedural imaging.
Diffusion Weighted MRI efficacy assessment. | Within 48 hours
  In case of DW-MRI evaluation, new ischemic lesions according to protocol criteria in postprocedural imaging.
Intravascular Ultrasound Stent Evaluation | Periprocedural
  In case of IVUS examination, postprocedural stent expansion, apposition and carotid plaque sequestration evaluation.
Ipsilateral Stroke incidence | From one month until one year after the procedure.
  Ischemic stoke at the site of index procedure.
Ipsilateral Stroke incidence | From one year until five years after the procedure.
  Ischemic stoke at the site of index procedure.
Any stroke incidence | Within five years from the procedure.
  Any stroke during study observational period.
Peak Systolic Velocity in Duplex Ultrasound evaluation in target vessel | Periprocedural
  Peak-systolic and End-diastolic Velocities assessed with DUS peri-proceduraly.
Peak Systolic Velocity in Duplex Ultrasound evaluation in target vessel | Within 30 days after index procedure.
  Peak-systolic and End-diastolic Velocities assessed with DUS 30 day after discharge.
Peak Systolic Velocity in Duplex Ultrasound evaluation in target vessel | One year after index procedure.
  Peak-systolic and End-diastolic Velocities assessed with DUS one year after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Musialek, MD, PhD, Principal Investigator — Jagiellonian University
Locations (1):
- Department of Cardiac and Vascular Diseases, The John Paul II Hospital, Krakow, Maloplska, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aboyans V, Ricco JB, Bartelink MEL, Bjorck M, Brodmann M, Cohnert T, Collet JP, Czerny M, De Carlo M, Debusa S, Espinola-Klein C, Kahan T, Kownator S, Mazzolai L, Naylora AR, Roffi M, Rotherb J, Sprynger M, Tendera M, Tepe G, Venermoa M, Vlachopoulos C, Desormais I. 2017 ESC Guidelines on the Diagnosis and Treatment of Peripheral Arterial Diseases, in collaboration with the European Society for Vascular Surgery (ESVS). Rev Esp Cardiol (Engl Ed). 2018 Feb;71(2):111. doi: 10.1016/j.rec.2017.12.014. No abstract available. English, Spanish. PMID 29425606
- [Background] Brott TG, Howard G, Roubin GS, Meschia JF, Mackey A, Brooks W, Moore WS, Hill MD, Mantese VA, Clark WM, Timaran CH, Heck D, Leimgruber PP, Sheffet AJ, Howard VJ, Chaturvedi S, Lal BK, Voeks JH, Hobson RW 2nd; CREST Investigators. Long-Term Results of Stenting versus Endarterectomy for Carotid-Artery Stenosis. N Engl J Med. 2016 Mar 17;374(11):1021-31. doi: 10.1056/NEJMoa1505215. Epub 2016 Feb 18. PMID 26890472
- [Background] Rosenfield K, Matsumura JS, Chaturvedi S, Riles T, Ansel GM, Metzger DC, Wechsler L, Jaff MR, Gray W; ACT I Investigators. Randomized Trial of Stent versus Surgery for Asymptomatic Carotid Stenosis. N Engl J Med. 2016 Mar 17;374(11):1011-20. doi: 10.1056/NEJMoa1515706. Epub 2016 Feb 17. PMID 26886419
- [Background] Sardar P, Chatterjee S, Aronow HD, Kundu A, Ramchand P, Mukherjee D, Nairooz R, Gray WA, White CJ, Jaff MR, Rosenfield K, Giri J. Carotid Artery Stenting Versus Endarterectomy for Stroke Prevention: A Meta-Analysis of Clinical Trials. J Am Coll Cardiol. 2017 May 9;69(18):2266-2275. doi: 10.1016/j.jacc.2017.02.053. PMID 28473130
- [Background] Janczak D, Malinowski M, Ziomek A, Kobecki J, Lesniak M, Dorobisz T, Dorobisz K, Janczak D, Chabowski M. Carotid artery stenting versus endarterectomy for the treatment of both symptomatic and asymptomatic patients with carotid artery stenosis: 2 years' experience in a high-volume center. Adv Clin Exp Med. 2018 Dec;27(12):1691-1695. doi: 10.17219/acem/75902. PMID 30063301
- [Background] de Donato G, Setacci F, Sirignano P, Galzerano G, Cappelli A, Setacci C. Optical coherence tomography after carotid stenting: rate of stent malapposition, plaque prolapse and fibrous cap rupture according to stent design. Eur J Vasc Endovasc Surg. 2013 Jun;45(6):579-87. doi: 10.1016/j.ejvs.2013.03.005. Epub 2013 Apr 10. PMID 23582886
- [Background] Kotsugi M, Takayama K, Myouchin K, Wada T, Nakagawa I, Nakagawa H, Taoka T, Kurokawa S, Nakase H, Kichikawa K. Carotid Artery Stenting: Investigation of Plaque Protrusion Incidence and Prognosis. JACC Cardiovasc Interv. 2017 Apr 24;10(8):824-831. doi: 10.1016/j.jcin.2017.01.029. PMID 28427600
- [Background] Schofer J, Musialek P, Bijuklic K, Kolvenbach R, Trystula M, Siudak Z, Sievert H. A Prospective, Multicenter Study of a Novel Mesh-Covered Carotid Stent: The CGuard CARENET Trial (Carotid Embolic Protection Using MicroNet). JACC Cardiovasc Interv. 2015 Aug 17;8(9):1229-1234. doi: 10.1016/j.jcin.2015.04.016. PMID 26292586
- [Background] Pieniazek P, Musialek P, Kablak-Ziembicka A, Tekieli L, Motyl R, Przewlocki T, Moczulski Z, Pasowicz M, Sokolowski A, Lesniak-Sobelga A, Zmudka K, Tracz W. Carotid artery stenting with patient- and lesion-tailored selection of the neuroprotection system and stent type: early and 5-year results from a prospective academic registry of 535 consecutive procedures (TARGET-CAS). J Endovasc Ther. 2008 Jun;15(3):249-62. doi: 10.1583/07-2264.1. PMID 18540694
- [Background] Musialek P, Grunwald IQ. How asymptomatic is "asymptomatic" carotid stenosis? Resolving fundamental confusion(s) - and confusions yet to be resolved. Pol Arch Intern Med. 2017 Nov 30;127(11):718-719. doi: 10.20452/pamw.4157. Epub 2017 Nov 30. No abstract available. PMID 29192895
- [Background] Musialek P, Hopf-Jensen S. Commentary: Carotid Artery Revascularization for Stroke Prevention: A New Era. J Endovasc Ther. 2017 Feb;24(1):138-148. doi: 10.1177/1526602816671263. Epub 2016 Oct 13. No abstract available. PMID 27733691
- [Background] Musialek P, Hopkins LN, Siddiqui AH. One swallow does not a summer make but many swallows do: accumulating clinical evidence for nearly-eliminated peri-procedural and 30-day complications with mesh-covered stents transforms the carotid revascularisation field. Postepy Kardiol Interwencyjnej. 2017;13(2):95-106. doi: 10.5114/pwki.2017.69012. Epub 2017 Jul 19. PMID 28798779
- [Background] Stabile E, de Donato G, Musialek P, De Loose K, Nerla R, Sirignano P, Chianese S, Mazurek A, Tesorio T, Bosiers M, Setacci C, Speziale F, Micari A, Esposito G. Use of Dual-Layered Stents in Endovascular Treatment of Extracranial Stenosis of the Internal Carotid Artery: Results of a Patient-Based Meta-Analysis of 4 Clinical Studies. JACC Cardiovasc Interv. 2018 Dec 10;11(23):2405-2411. doi: 10.1016/j.jcin.2018.06.047. PMID 30522670
- [Background] Musialek P. TASTE-less endpoint of 30-day mortality (and some other issues with TASTE) in evaluating the effectiveness of thrombus aspiration in STEMI: not the "evidence" to change the current practice of routine consideration of manual thrombus extraction. Kardiol Pol. 2014;72(6):479-87. doi: 10.5603/KP.a2014.0022. Epub 2014 Feb 14. No abstract available. PMID 24526550
- [Result] Musialek P, Mazurek A, Trystula M, Borratynska A, Lesniak-Sobelga A, Urbanczyk M, Banys RP, Brzychczy A, Zajdel W, Partyka L, Zmudka K, Podolec P. Novel PARADIGM in carotid revascularisation: Prospective evaluation of All-comer peRcutaneous cArotiD revascularisation in symptomatic and Increased-risk asymptomatic carotid artery stenosis using CGuard MicroNet-covered embolic prevention stent system. EuroIntervention. 2016 Aug 5;12(5):e658-70. doi: 10.4244/EIJY16M05_02. PMID 27180302